CLINICAL TRIAL: NCT04907786
Title: Coronary Computed Tomography Angiography Guidance in Invasive Coronary Angiography; a Prospective Registry Study
Brief Title: CCTA-guided Ultraselective Invasive Coronary Angiography
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Collaborators: The Elisabeth-TweeSteden Hospital (Other)
Responsible Party: Principal Investigator, Lokien van Nunen, Principal Investigator, Catharina Ziekenhuis Eindhoven
Other Study IDs: Ultraselective Registry
Record Dates: First submitted 2021-05-21; First posted 2021-06-01 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Coronary Artery Disease
Keywords: Invasive coronary angiography; Coronary computed tomographic angiography; Radiation exposure; Contrast volume; Procedure costs
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study population: All patients eligible for participation in this registry are aged 18-80 years old and undergoing invasive coronary angiography because of abnormalities found on CCTA in either the left or right coronary artery and no or minimal stenosis (CAD-RADS 0-1; 0-24% stenosis) in the contralateral coronary artery. Patients will be asked for written informed consent to register their clinical data in an anonymized database. The period between CCTA and ICA may not exceed 90 days, in order to prevent possible aggravation of coronary artery disease between both examinations.

SUMMARY:
Coronary artery disease (CAD) is the leading cause of death in adults in the United States.[1] In the latest guidelines of the European Society of Cardiology anatomical non-invasive imaging by coronary computed tomography angiography (CCTA) plays an important role in the diagnosis of the presence of CAD in patients without a history of CAD and a low to intermediate likelihood.[2] CCTA provides high accuracy for the detection of coronary artery disease by visualizing the coronary artery lumen using an intravenous contrast agent.[3] However to determine the hemodynamical significance of CCTA-identified stenosis, invasive coronary angiography (ICA) with or without functional testing is still required. [4] During the ICA as per protocol the complete coronary artery system is visualized again. In patients with abnormalities on CCTA in only one coronary artery, i.e. only the left coronary artery (LCA) or the right coronary artery (RCA), the ICA procedure might be simplified by 'ultraselectively' visualizing only the coronary artery of interest and refraining from angiographic visualization of the contralateral coronary artery without abnormalities on CCTA (with an excellent negative predictive value of 95-99%).[5-7] Such an ultraselective strategy might reduce procedure time, usage of catheters, complication risk and the amount of contrast agent and radiation exposure.

A recent retrospective study in three hospitals in the Netherlands showed CCTA to be extremely accurate in predicting a normal contralateral coronary artery in patients with coronary artery disease limited to the left or right coronary artery. Therefore, a CCTA-guided ultraselective ICA approach would have been safe and feasible and would have led to a considerable decrease in procedure time and radiation exposure.

However, the analysis was hampered by the retrospective design. The potential benefits in salvage of procedure time and radiation exposure might be overestimated and it turned out to be impossible to measure the effects on contrast use, catheter use and procedure costs. Moreover, in the retrospective study only a small portion of the study population had abnormalities in the right coronary artery, thereby questioning the results of this study to safely be extrapolated to this category of patients with abnormalities in the RCA.

This dual-center prospective registry study is designed to answer these remaining questions and to further investigate the potential benefit of an ultraselective ICA approach.

DETAILED DESCRIPTION:
Study design & patient population

The study is a dual-center prospective registry in two hospitals in the Netherlands. All patients eligible for participation in this registry are aged 18-80 years old and undergoing invasive coronary angiography because of abnormalities found on CCTA in either the left or right coronary artery and no or minimal stenosis (CAD-RADS 0-1; 0-24% stenosis) in the contralateral coronary artery.

Patients will be asked for written informed consent to register their clinical data in an anonymized database. The period between CCTA and ICA may not exceed 90 days, in order to prevent possible aggravation of coronary artery disease between both examinations.

Clinical characteristics (age, gender, risk factors, relevant medical history) and CCTA data will be included in the database. All procedural characteristics and findings of the invasive coronary angiography procedure will be logged, including access site, procedural planning (which coronary artery to be visualized first), procedure duration, amount and type of catheters used, amount of radiation exposure and contrast volume, procedural findings, type of coronary intervention (if applicable), and complications. Procedure duration is defined as the time needed for the diagnostic part of the ICA procedure, possible further functional invasive testing and/or percutaneous coronary intervention is excluded. ICA data will be compared to the CCTA data on a per-patient level. No further follow-up is planned after the invasive coronary angiography with regards to participating in this registry.

Informed consent

If patients provide informed consent, the data will be registered in an anonymized database. Patients can withdraw from this study at any time at their own request, or they may be withdrawn at the discretion of the investigator for behavioral, or administrative reasons. The reason(s) for discontinuation will be documented and may include: the subject voluntarily withdraws from registry.

Since the patients will not be subjected to any additional procedures, rules or behavior and the data will be anonymized, we believe this research design does not fall under the scope of the Medical Research Involving Human Subjects Act (WMO).

Database and data protection

Data will be stored anonymized in an online database and will only be accessible to the involved researchers. Personal data will comply to the Dutch Personal Data Protection Act. Site investigators will only be able to add patients from their own site, and will only be able to see patients from their own site. Data generated will be encoded and a separate patient identification log will be created for each site, and stored at each site separately. The key to the code will be available to specific site investigators only. There will be at least one study coordinator that has access to all records of all sites. In the future data from other centers could be included into the database using this similar pattern to ensure data protection.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing invasive coronary angiography because of abnormalities found on CCTA in either the left or right coronary artery and no or minimal stenosis (CAD-RADS 0-1; 0-24% stenosis) in the contralateral coronary artery within 90 days.

Exclusion Criteria:

* Refusal of informed consent
* Abnormalities in both coronary arteries on CCTA
* Prior PCI
* Prior coronary artery bypass grafting (CABG)
* Major allergy to iodinated contrast agent
* Inability to provide informed consent, and/or known pregnancy.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The prospected study population is 250 patients. This study population allows for enough statistical power to answer all endpoints as described above. Due to the fact that only a few patients with abnormalities on the CCTA limited to the RCA were analyzed in the retrospective study, we defined that at least 15% of the patient population must consist of patients with an abnormal RCA on CCTA. In order to reach this distribution, inclusion of patients with abnormalities in the LCA on CCTA may be halted in favor of patients with abnormalities in the RCA.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of CCTA | At the end of the invasive coronary angiography procedure, an average of 25 minutes
  The accuracy of CCTA to defer invasive angiography of the contralateral coronary artery, in patients with abnormalities on CCTA limited to either the left or right coronary artery and a normal or minimal abnormal contralateral artery (defined as CAD-RADS 0-1; 0-24% stenosis)

SECONDARY OUTCOMES:
Reduction in procedure time | At the end of the invasive coronary angiography procedure, an average of 25 minutes.
  The time to visualize the contralateral coronary artery without abnormalities on CCTA will be considered as superfluous and is therefore a potential benefit of an ultraselective ICA.
Reduction in radiation | At the end of the invasive coronary angiography procedure, an average of 25 minutes
  The radiation used to to visualize the contralateral coronary artery without abnormalities on CCTA will will be considered as superfluous and is therefore a potential benefit of an ultraselective ICA.
Reduction in contrast volume | At the end of the invasive coronary angiography procedure, an average of 25 minutes
  The contrast volume used to to visualize the contralateral coronary artery without abnormalities on CCTA will be considered as superfluous and is therefore a potential benefit of an ultraselective ICA.
Reduction in catheter usage | At the end of the invasive coronary angiography procedure, an average of 25 minutes
  The amount of catheter used to visualize the contralateral coronary artery without abnormalities on CCTA will be considered as superfluous and is therefore a potential benefit of an ultraselective ICA.

CONTACTS AND LOCATIONS:
Locations (1):
- Catharina Hospital, Eindhoven, North Brabant, Netherlands

REFERENCES:
- [Background] Benjamin EJ, Virani SS, Callaway CW, Chamberlain AM, Chang AR, Cheng S, Chiuve SE, Cushman M, Delling FN, Deo R, de Ferranti SD, Ferguson JF, Fornage M, Gillespie C, Isasi CR, Jimenez MC, Jordan LC, Judd SE, Lackland D, Lichtman JH, Lisabeth L, Liu S, Longenecker CT, Lutsey PL, Mackey JS, Matchar DB, Matsushita K, Mussolino ME, Nasir K, O'Flaherty M, Palaniappan LP, Pandey A, Pandey DK, Reeves MJ, Ritchey MD, Rodriguez CJ, Roth GA, Rosamond WD, Sampson UKA, Satou GM, Shah SH, Spartano NL, Tirschwell DL, Tsao CW, Voeks JH, Willey JZ, Wilkins JT, Wu JH, Alger HM, Wong SS, Muntner P; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2018 Update: A Report From the American Heart Association. Circulation. 2018 Mar 20;137(12):e67-e492. doi: 10.1161/CIR.0000000000000558. Epub 2018 Jan 31. No abstract available. PMID 29386200
- [Background] Knuuti J, Wijns W, Saraste A, Capodanno D, Barbato E, Funck-Brentano C, Prescott E, Storey RF, Deaton C, Cuisset T, Agewall S, Dickstein K, Edvardsen T, Escaned J, Gersh BJ, Svitil P, Gilard M, Hasdai D, Hatala R, Mahfoud F, Masip J, Muneretto C, Valgimigli M, Achenbach S, Bax JJ; ESC Scientific Document Group. 2019 ESC Guidelines for the diagnosis and management of chronic coronary syndromes. Eur Heart J. 2020 Jan 14;41(3):407-477. doi: 10.1093/eurheartj/ehz425. No abstract available. PMID 31504439
- [Background] Knuuti J, Ballo H, Juarez-Orozco LE, Saraste A, Kolh P, Rutjes AWS, Juni P, Windecker S, Bax JJ, Wijns W. The performance of non-invasive tests to rule-in and rule-out significant coronary artery stenosis in patients with stable angina: a meta-analysis focused on post-test disease probability. Eur Heart J. 2018 Sep 14;39(35):3322-3330. doi: 10.1093/eurheartj/ehy267. PMID 29850808
- [Background] Tonino PA, Fearon WF, De Bruyne B, Oldroyd KG, Leesar MA, Ver Lee PN, Maccarthy PA, Van't Veer M, Pijls NH. Angiographic versus functional severity of coronary artery stenoses in the FAME study fractional flow reserve versus angiography in multivessel evaluation. J Am Coll Cardiol. 2010 Jun 22;55(25):2816-21. doi: 10.1016/j.jacc.2009.11.096. PMID 20579537
- [Background] Budoff MJ, Dowe D, Jollis JG, Gitter M, Sutherland J, Halamert E, Scherer M, Bellinger R, Martin A, Benton R, Delago A, Min JK. Diagnostic performance of 64-multidetector row coronary computed tomographic angiography for evaluation of coronary artery stenosis in individuals without known coronary artery disease: results from the prospective multicenter ACCURACY (Assessment by Coronary Computed Tomographic Angiography of Individuals Undergoing Invasive Coronary Angiography) trial. J Am Coll Cardiol. 2008 Nov 18;52(21):1724-32. doi: 10.1016/j.jacc.2008.07.031. PMID 19007693
- [Background] Meijboom WB, Meijs MF, Schuijf JD, Cramer MJ, Mollet NR, van Mieghem CA, Nieman K, van Werkhoven JM, Pundziute G, Weustink AC, de Vos AM, Pugliese F, Rensing B, Jukema JW, Bax JJ, Prokop M, Doevendans PA, Hunink MG, Krestin GP, de Feyter PJ. Diagnostic accuracy of 64-slice computed tomography coronary angiography: a prospective, multicenter, multivendor study. J Am Coll Cardiol. 2008 Dec 16;52(25):2135-44. doi: 10.1016/j.jacc.2008.08.058. PMID 19095130
- [Background] Miller JM, Rochitte CE, Dewey M, Arbab-Zadeh A, Niinuma H, Gottlieb I, Paul N, Clouse ME, Shapiro EP, Hoe J, Lardo AC, Bush DE, de Roos A, Cox C, Brinker J, Lima JA. Diagnostic performance of coronary angiography by 64-row CT. N Engl J Med. 2008 Nov 27;359(22):2324-36. doi: 10.1056/NEJMoa0806576. PMID 19038879